CLINICAL TRIAL: NCT05373719
Title: Endpoint Enabling Study of Cyclin-dependent Kinase-like 5 (CDKL5) Deficiency Disorder (CDD)
Brief Title: Observational Study in Patients With Cyclin-dependent Kinase-like 5 Deficiency Disorder
Acronym: CANDID
Status: Active, not recruiting | Type: Observational
Sponsor: Loulou Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LLF001
Record Dates: First submitted 2022-05-06; First posted 2022-05-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cyclin-Dependent Kinase-Like 5 Deficiency Disorder
Keywords: Cyclin-Dependent Kinase-Like 5 Deficiency Disorder; CDKL5; CDD
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- 0-2 Years of Age: Patients from birth to 2 years of age at time of study entry
  Interventions: Other: No intervention; observational
- 3-5 Years of Age: Patients aged 3 to 5 years at time of study entry
  Interventions: Other: No intervention; observational
- 6-12 Years of Age: Patients aged 6 to 12 years at time of study entry
  Interventions: Other: No intervention; observational
- 13-55 Years of Age: Patients aged 13 to 55 years at time of study entry
  Interventions: Other: No intervention; observational

INTERVENTIONS:
Other: No intervention; observational — No intervention; observational

SUMMARY:
Observational, noninterventional, 3-year study to examine the presence of detectable differences in neurocognitive, developmental, motor, neurophysiologic, and quality of life measures over time in patients with cyclin-dependent kinase-like 5 deficiency disorder.

DETAILED DESCRIPTION:
This is an observational study to examine the presence of detectable differences in neurocognitive, developmental, motor, neurophysiologic, and quality of life measures over time in approximately up to 100 patients aged birth to 55 years and diagnosed with cyclin-dependent kinase-like 5 deficiency disorder. Operational performance across age groups and languages will be assessed throughout the study, and Baseline cohort characteristics will be assessed throughout enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of Cyclin-dependent Kinase-like 5 (CDKL5) deficiency disorder with pathogenic or likely pathogenic of CDKL5 variants
2. Ages newborn to 55 years old
3. Parent/Caregiver who is willing and capable of providing written informed consent
4. Parent/caregiver lives with or has daily contact with study participant and able to provide consistent information across the study

Exclusion Criteria:

1. Any clinically significant neurocognitive deficit not attributable to Cyclin-dependent Kinase-like 5 (CDKL5) deficiency disorder or a secondary cause that may, in the opinion of the investigator, confound interpretation of study results (e.g., extreme prematurity, other genetic variants, unclassified CDKL5 variant, abnormal brain imaging, imaging and/or injury not otherwise attributable to CDD).
2. Any condition that, in the opinion of the investigator, would put the patient at undue risk or make it unsafe for the patient to participate
3. Any condition which would make the individual or the caregiver, in the opinion of the investigator, unsuitable for the study

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a multi-center study to be conducted in multiple countries. The study will enroll patients diagnosed with Cyclin-dependent Kinase-like 5 (CDKL5) deficiency disorder, from birth to 55 years of age, at a participating site.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Bayley Scale of Infant and Toddler Development, Fourth Edition (BSID-4) | Baseline
  Suitability of this cognition and global development scale in CDD will be assessed based on the number of tests completed, ceiling/floor effect and variance estimate.
Vineland 3 | Baseline
  Suitability of this adaptive behavior scale in CDD will be assessed based on the number of tests completed, ceiling/floor effect and variance estimate.
Gross Motor Function Measure (GMFM) | Baseline
  Suitability of this motor function scale in CDD will be assessed based on the number of tests completed, ceiling/floor effect and variance estimate.
Sleep Disturbance Scale for Children (SDSC) | Baseline
  Suitability of this sleep quality scale in CDD will be assessed based on the number of tests completed, ceiling/floor effect and variance estimate.

SECONDARY OUTCOMES:
Changes in test results over time. | 36 months
Correlations between age and test results. | 36 months
Correlations between gender and test results. | 36 months
Correlation between test results and seizure severity. | 36 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (9):
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - New York University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Childrens Hospital of Philadlephia Division of Neurology, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - Alberta Children's Hospital, Pediatric Epilepsy and Child Neurology, Calgary
  - The Hospital of Sick Children, Toronto
- Hopital Necker- Enfants Malades, Paris, France
- Germany (2):
  - DRK Berlin - Epilepsiezentrum und Neuropädiatrie, Berlin
  - Schön Klinik Vogtareuth, Vogtareuth
- Italy (4):
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Fondazione Policlinico Universitario A Gemelli, IRCCS, Roma
  - Ospedale Pediatrico Bambino Gesù, Rome
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Spain (3):
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Ruber Internacional Hospital, Madrid
  - Hospital UniversitarioVithas Madrid, Madrid
- Mediclinic, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes